CLINICAL TRIAL: NCT05190913
Title: The Effect of Instrumented and Non-Instrumental Perineal Massage on Birth Results in the Active Phase of Labor
Brief Title: Instrumental and Non-Instrumental Perineal Message and Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Meryem Metinoglu, Lecturer, Namik Kemal University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: TNKU-M.Metinoglu-001
Record Dates: First submitted 2021-12-04; First posted 2022-01-13 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Labor
Keywords: Labor Pain; Episiotomy; birth satisfaction; birth
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: Intervention I group (n:40) from two different experimental groups will be given instrumental perineal massage, and intervention II group (n:40) from the other experimental group will be given non-instrumental perineal massage. No intervention is planned for the control group (n:40).
Who Masked: Outcomes Assessor
Masking Description: Due to the design of the study, single or double masking cannot be done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initiative group I (Experimental): In the active phase of labor, perineal massage will be performed with the device at an interval of one hour.
  Interventions: Other: Instrumental perineal massage
- Initiative group II (Experimental): During the active phase of labor, manual perineal massage will be performed with an interval of one hour.
  Interventions: Other: manual perineal massage

INTERVENTIONS:
Other: Instrumental perineal massage — In the active phase of labor, perineal massage will be performed with an instrument twice with an interval of one hour.
  Arms: Initiative group I
Other: manual perineal massage — In the active phase of labor, manual perineal massage is performed twice an hour apart.
  Arms: Initiative group II

SUMMARY:
Today, the increase in the costs of applications in the health care system makes it difficult for easy and inexpensive methods to be used based on evidence. In this study, the episiotomy rate, episiotomy length, perineal pain at birth and postpartum period, perineal trauma, newborn 1st min. and 5 min. It was planned as a Randomized Controlled Experimental study to examine the effect of APGAR score on birth outcomes such as the duration of the first and second stages of labor and birth satisfaction.

The universe of the research was carried out between December 2021-2022 in University Hospital and City Hospital Pregnant women at 38-42 weeks of gestation who are admitted to the maternity ward to give birth. Power analysis was performed using the GPower program in order to sample size. In determining the sample size, the article titled "The Effect of Perineal Massage During Labor in Nulliparous Women on Birth Comfort, Perineal Pain and Trauma" (Yaşar, 2019) was used. Considering the total mean scores of the GCS scale in intervention and control groups, Type 1 error amount was 0.01, test power was 0.99, and effect size was 1.1276841; The minimum required sample size was determined as 80 (40 interventions + 40 control groups) for the intervention and control groups. In line with these data, it was decided that the sample size would be 120 pregnant women who agreed to be in the study and met the inclusion criteria, 40 in the intervention-1 group to be given instrumental perineal massage, 40 in the intervention-2 group that would receive non-instrumental perineal massage, and 40 in the control group.

Frequency and mean values will be used in the evaluation of descriptive data, and independent sample t-test, chi-square test, fisher chi-square test and ANOVA will be used in the analysis of data showing normal distribution. The Mann Whitney U test is planned to be used in the analysis of data that do not show normal distribution. Normal distribution in the analysis of the relationship between prenatal instrument perineal massage and GCS scores, quality of pain, length of episiotomy, condition of the perineal region, duration of the first and second stages of labor, total delivery time, APGAR 1st and 5th minute scores, and parameters related to postpartum satisfaction Pearson correlation test will be used. All the results will be evaluated at the 95% confidence interval, at the 0.05 significance level.

DETAILED DESCRIPTION:
Randomization: In order to prevent the women in the intervention and control groups from being influenced by each other, a random selection was made between the two hospitals where the study would be conducted by drawing lots. According to this election, Tekirdag Dr. The women who will be included in the study from İsmail Fehmi Cumalıoğlu City Hospital will be included in the control group, and the women from the Tekirdağ Namık Kemal University Hospital will be included in the Intervention 1 and Interference 2 groups. Pregnant women to be sampled within intervention 1, intervention 2 and control groups will be determined by systematic random sampling method, one of the probabilistic sampling methods. The distribution within the group was made with a simple random selection method using the computer program module (https://www.calculatorsoup.com/calculators/statistics/random-number-generator.php). According to these results, the pregnant women to be included in the group are listed below in order of admission to the hospital.

Intervention Group 1 (Instrumental perineal massage group); Between October 2020 and March 2021, 86 women had normal vaginal deliveries in the obstetrics clinic of Tekirdağ Namık Kemal University Hospital. In this study, which was planned with reference to this number, the number of pregnant women to be included in the intervention1 group was made using a simple random selection method using the computer program module (https://www.calculatorsoup.com/calculators/statistics/random-number-generator.php). The order of application to the intervention 1 group 1. 4. 5. 8. 11. 14. 16. 20. 21. 23. 24. 25. 28. 29. 33. 34. 35. 39. 40. 43. 44. 46. 47 Pregnant women who are 52. 53. 56. 58. 59. 63. 64. 65. 70. 71. 72. 75. 76. 79. 82. 83. 86. will be taken.

Intervention Group 2 (The group that will receive manual perineal massage); Between October 2020 and March 2021, 86 women delivered vaginally to Tekirdağ Namık Kemal University Hospital's obstetrics clinic. In this study, which was planned with reference to this number, the number of pregnant women to be included in the intervention 2 group was made using a simple random selection method by using the computer program module (https://www.calculatorsoup.com/calculators/statistics/random-number-generator.php). The order of application to the initiative 2 group 2. 3. 6. 7. 9. 10. 12. 13. 15.17. 18. 19. 22. 27. 30. 31. 32. 36. 38. 41. 42. 45. 48. 49. 51. 54. 55. 60. 61. 66. 67. 68. 69. 73. 74. Pregnant women who are 77. 78. 80. 81. 85. will be accepted. The pregnant woman who was excluded from the study due to any of the reasons stated in the randomization will be replaced by the pregnant who was admitted for the next delivery and her sequence number will be given to the next pregnant woman.

Control Group; Tekirdag Dr. Between October 2020 and March 2021, 252 women delivered vaginally to İsmail Fehmi Cumalıoğlu City Hospital's maternity clinic. In this study, which was planned with reference to this number, the number of pregnant women to be included in the control group was made using a simple random selection method using the computer program module (https://www.calculatorsoup.com/calculators/statistics/random-number-generator.php). Tekirdag Dr. to the control group. The order of application to İsmail Fehmi Cumalıoğlu City Hospital as of October 2021 is 9 15 18 20 34 43 44 46 49 53 60 64 65 67 77 78 81 84 102 103 108 118 120 128 131 136 152 158 163 171 178 179 184 186 187 198 205 206 228 230 pregnant women will be taken.

If the hospital in the intervention and control groups receives the news that there is a pregnant hospitalization meeting the inclusion criteria at the same time, the pregnant women in this center will be given priority, since the number of births in the hospital planned to be included in the intervention group is lower.

Data Collection Method: The application steps of the study are given below. Stage 1: A preliminary application will be made in the research, and the intelligibility, applicability and total application times of the forms/scales to be used in data collection will be evaluated. The pre-application is planned to be done on five pregnant women and it is planned to determine the problems in understanding the questions in the forms in line with the feedback. Among the women in both the intervention and control groups, the pregnant women who met the sampling criteria but did not accept the study or were taken to the cesarean section after accepting the study will be excluded from the study. The pregnant who had to be canceled due to any of the reasons stated in the randomization will be replaced by the pregnant hospitalized for the next delivery, and the targeted number of pregnant women will be reached by giving the next pregnant woman's sequence number. Determination of groups by randomization and obtaining their consent will be carried out at this stage. Personal Information Form, Labor Evaluation Form Part I, Visual Comparison Scale (GCS) will be applied to all pregnant women divided into groups in the latent phase of the first stage of labor.

Stage 2: Instrumental perineal massage will be applied to the Interference-1 group, whose cervical opening is 4-8 cm and is in the active phase of labor. Materials to be used: Perineum massage device (EPİ-NO) is a water-based lubricant. The process will be applied in 10 minutes, with two applications from the active phase to the transition phase and an average of one hour break after each application . Perineal massage will be performed at the same time intervals and for the same durations for the Initiative-2 Group, which receives manual perineal massage. Perineum massage will not be given to the control group pregnant women, and routine delivery room practices will be continued by the service workers. At this stage, the pregnant women are given the Labor Evaluation Form II. Section and GLO will be applied.

3. Stage: It is the stage where the transitional phase of the pregnant women divided into groups is completed and the births take place. For all three groups, there was no other treatment except clinical routine applications.

Stage 4: Within the first 48 hours of postpartum postpartum, Labor Evaluation Form III. It will be watched with the Chapter . If analgesia and local anesthesia are applied, it will be expected that the effect will wear off, and six hours after the second stage of labor, the puerperant women will be asked to mark the perineal pain level on the VCO visual. REEDA Scale will be used for the evaluation of the perineal area (Episiotomy, pole, tear).

5th Stage: After confirming that no analgesic was used at least six hours before the postpartum was called by phone on the 10th day of postpartum, GCS for perineal pain level, REEDA Scale to evaluate the condition of the perineal area, and DME to assess satisfaction at birth. Data will be collected by querying with.

Materials to be used in the research: Perineal massage device (EPİ-NO), water-based lubricant.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* No vision and hearing problems
* At least primary school graduate and no language problems
* Those between the ages of 18-35
* 38th-42nd of pregnancy. in the week
* Does not feel uncomfortable being touched by the genital area
* Those who are willing to have a normal delivery and have a vaginal delivery indication
* During the first stage of labor, analgesia and anesthesia are not used.
* Head presenter
* Single pregnancy
* Those who do not have a risky pregnancy (Dystosiler, Presanta previa, threat of premature birth, premature rupture of membranes, preeclampsia, eclampsia, hyperemesis gravidarum, ablatio placenta, placenta accreta, intrauterine growth retardation, cord anomaly, vaginal bleeding, etc.)

Exclusion Criteria:

* Non-Turkish citizens
* Planned cesarean section
* Having genital infection
* A different perineal massager
* Pregnant women with narcotic and analgesic addiction and who were administered narcotic analgesics during the data collection process.
* Known chronic disease (heart disease, hypertension, diabetes, kidney disease, etc.) systemic disease
* Having a neurological disease
* Non-pharmacological pain control methods at birth (respiratory exercise techniques, massage, intradermal water injection, relaxation and relaxation methods, mental/mental stimulation, Transcutaneous electrical nerve stimulation, etc.). using.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Labor Evaluation Form Part I | The progression time of vaginal dilatation at birth may vary from person to person. For this reason, the questionnaire will be applied at the beginning of the birth process, before the vaginal dilatation is 4 cm.
  I. It will be applied in the latent phase of labor (cervical dilatation: 0-4 cm).
  II.It will be applied in the active phase of labor (cervical dilatation: 4-8 cm).
  III.Until two days after birth
Visual analog scale | The progression time of vaginal dilatation at birth may vary from person to person. For this reason, the questionnaire will be applied at the beginning of the birth process, before the vaginal dilatation is 4 cm.
  Birth pain. VAS is a horizontal or vertical line of 10 cm/100 mm that starts with "No pain" and ends with "Unbearable pain." No pain is written on one end and very severe or unbearable pain is written on the other end on the scale during the measurement and the patient marks their current state on this line. The length of the distance from no pain to the point marked by the patient indicates the patient's pain.
Labor Evaluation Form Part II | The progression time of vaginal dilatation at birth may vary from person to person. For this reason, the questionnaire will be applied at the beginning of the birth process, before the vaginal dilatation is 8 cm.
  It will be applied during the active period of labor (cervical dilatation: 5-8 cm).
  II.It will be applied in the active phase of labor (cervical dilatation: 4-8 cm).
  III.Until two days after birth
Labor Evaluation Form Part III | This form is evaluated within 48 hours of postpartum
  It will be applied within the first 48 hours after the birth is completed.
REEDA Scale | The REEDA score is evaluated in the 48th hour after delivery.
  This scale includes five factors that indicate perineal wound healing. These; These are redness (redness), edema (edema), ecchymosis (ecchymosis), discharge (discharge), approximation (approaching wound ends). Each factor takes values between 0-3. A total REEDA score (0-15) is obtained by evaluating these five improvement factors. The lowest score is 0 points, the highest score is 15 points. Higher scores indicate more tissue trauma.
Birth satisfaction scale | This form is evaluated postpartum 10th day.
  The original of the scale used to evaluate women's perceptions of birth satisfaction is 30 items and is a five-point Likert type. It consists of 3 main themes: quality of care, personal characteristics of women and stress experienced during childbirth. A minimum of 30 and a maximum of 150 points can be obtained from the scale. The higher the score, the higher the level of satisfaction.
Visual analog scale | The VAS is evaluated postpartum10th day.
  It is a scale used to evaluate the severity of pain. participants are asked to mark or say the point on the line numbered from zero to 10 that corresponds to the pain.Zero points; While expressing no pain, 10 points indicates the most severe pain experienced.

SECONDARY OUTCOMES:
Visual analog scale | The progression time of vaginal dilatation at birth may vary from person to person. For this reason, the questionnaire will be applied at the beginning of the birth process, before the vaginal dilatation is 8 cm.
  Birth pain. VAS is a horizontal or vertical line of 10 cm/100 mm that starts with "No pain" and ends with "Unbearable pain." No pain is written on one end and very severe or unbearable pain is written on the other end on the scale during the measurement and the patient marks their current state on this line. The length of the distance from no pain to the point marked by the patient indicates the patient's pain.
Visual analog scale | The VAS is evaluated within 48 hours of postpartum after delivery
  Birth pain. VAS is a horizontal or vertical line of 10 cm/100 mm that starts with "No pain" and ends with "Unbearable pain." No pain is written on one end and very severe or unbearable pain is written on the other end on the scale during the measurement and the patient marks their current state on this line. The length of the distance from no pain to the point marked by the patient indicates the patient's pain.
REEDA Scale | The REEDA score is evaluated in the postpartum 10th day after delivery.
  This scale includes five factors that indicate perineal wound healing. These; These are redness (redness), edema (edema), ecchymosis (ecchymosis), discharge (discharge), approximation (approaching wound ends). Each factor takes values between 0-3. A total REEDA score (0-15) is obtained by evaluating these five improvement factors. The lowest score is 0 points, the highest score is 15 points. Higher scores indicate more tissue trauma.

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Metinoğlu, Principal Investigator — TNKU
Locations (1):
- Meryem Metinoğlu, Tekirdağ, Süleymanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdelhakim AM, Eldesouky E, Elmagd IA, Mohammed A, Farag EA, Mohammed AE, Hamam KM, Hussein AS, Ali AS, Keshta NHA, Hamza M, Samy A, Abdel-Latif AA. Antenatal perineal massage benefits in reducing perineal trauma and postpartum morbidities: a systematic review and meta-analysis of randomized controlled trials. Int Urogynecol J. 2020 Sep;31(9):1735-1745. doi: 10.1007/s00192-020-04302-8. Epub 2020 May 12. PMID 32399905
- [Background] Dencker A, Nilsson C, Begley C, Jangsten E, Mollberg M, Patel H, Wigert H, Hessman E, Sjoblom H, Sparud-Lundin C. Causes and outcomes in studies of fear of childbirth: A systematic review. Women Birth. 2019 Apr;32(2):99-111. doi: 10.1016/j.wombi.2018.07.004. Epub 2018 Aug 14. PMID 30115515
- [Background] Jahani Shoorab N, Mirteimouri M, Taghipour A, Latifnejad Roudsari R. Women's Experiences of Emotional Recovery from Childbirth-Related Perineal Trauma: A Qualitative Content Analysis. Int J Community Based Nurs Midwifery. 2019 Jul;7(3):181-191. doi: 10.30476/IJCBNM.2019.44993. PMID 31341917
- [Background] O'Connell MA, Khashan AS, Leahy-Warren P, Stewart F, O'Neill SM. Interventions for fear of childbirth including tocophobia. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013321. doi: 10.1002/14651858.CD013321.pub2. PMID 34231203
- [Background] Manresa M, Pereda A, Bataller E, Terre-Rull C, Ismail KM, Webb SS. Incidence of perineal pain and dyspareunia following spontaneous vaginal birth: a systematic review and meta-analysis. Int Urogynecol J. 2019 Jun;30(6):853-868. doi: 10.1007/s00192-019-03894-0. Epub 2019 Feb 15. PMID 30770967
- [Background] Kavvadias T, Hoesli I. The EpiNo(R) Device: Efficacy, Tolerability, and Impact on Pelvic Floor-Implications for Future Research. Obstet Gynecol Int. 2016;2016:3818240. doi: 10.1155/2016/3818240. Epub 2016 Feb 14. PMID 26981126
- [Background] Martin CH, Fleming V. The birth satisfaction scale. Int J Health Care Qual Assur. 2011;24(2):124-35. doi: 10.1108/09526861111105086. PMID 21456488
- [Background] Demsar K, Svetina M, Verdenik I, Tul N, Blickstein I, Globevnik Velikonja V. Tokophobia (fear of childbirth): prevalence and risk factors. J Perinat Med. 2018 Feb 23;46(2):151-154. doi: 10.1515/jpm-2016-0282. PMID 28379837
- See also: pubmed 32399905 — https://pubmed.ncbi.nlm.nih.gov/32399905/
- See also: pubmed 30115515 — https://pubmed.ncbi.nlm.nih.gov/30115515/
- See also: pubmed 31341917 — https://pubmed.ncbi.nlm.nih.gov/31341917/
- See also: pubmed 34231203 — https://pubmed.ncbi.nlm.nih.gov/34231203/
- See also: pubmed 30770967 — https://pubmed.ncbi.nlm.nih.gov/30770967/
- See also: pubmed 26981126 — https://pubmed.ncbi.nlm.nih.gov/26981126/
- See also: pubmed 21456488 — https://pubmed.ncbi.nlm.nih.gov/21456488/
- See also: pubmed 28379837 — https://pubmed.ncbi.nlm.nih.gov/28379837/
- See also: random number generator — http://clinicaltrials.gov
- See also: Referenced article for Gpower — http://abakus.inonu.edu.tr/xmlui/handle/11616/15104